CLINICAL TRIAL: NCT01198431
Title: Effects of Impaired Sleep on Energy Balance: A Randomized, 2-Condition, Crossover Study in Adolescents
Brief Title: Effects of Impaired Sleep on Energy Balance
Acronym: SLOPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Arne Astrup, Department of Human Nutrition, Faculty of LIFE Sciences, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OPUS-B261
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2010-09

CONDITIONS: Obesity; Sleep
Keywords: Appetite regulation; Physical activity; Energy balance
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Sleep Duration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep restriction (Experimental): Each participant will be engaged in three consecutive nights of 4 hours of sleep per night (from 3.00 a.m. to 7.00 a.m.)
  Interventions: Behavioral: Sleep duration
- Normal sleep duration (Placebo Comparator): Each participant will be engaged in three consecutive nights of 9 hours of sleep per night (from 10.00 p.m. to 7.00 a.m.)
  Interventions: Behavioral: Sleep duration

INTERVENTIONS:
Behavioral: Sleep duration — Duration of sleep per night
  Other Names: Sleep curtailment, acute sleep deprivation

SUMMARY:
The main aim of this study is to examine the effects of restricted sleep on energy and substrate metabolism as well as relevant hormonal systems that might be involved in the underlying mechanisms.

The investigators hypothesize that short-term sleep curtailment in adolescents is accompanied by 1) increased hunger and desire to eat; 2) increased spontaneous energy intake; 3) reduced spontaneous physical activity; and 4) increased fluctuation in hormones in a way that could favour a positive energy balance and potentially weight gain on the long run.

DETAILED DESCRIPTION:
The background for this project is that despite considerable knowledge of the mechanisms regulating body weight, the prevalence of obesity has not declined. The individual and environmental factors that play a part in energy balance are still not completely understood, and current methods for loosing and maintaining body weight are generally unsuccessful. Knowledge about what brings about changes in metabolism and lifestyle is lacking.

Reduced sleep duration has been observed in parallel with increases in body weight. Lack of sleep has become a hallmark of modern man, and both children and adults sleep less today than just a few decades ago. Research suggests that both too much and too little sleep can lead to obesity, but correlations between sleep deprivation and other lifestyle-related ailments have also been observed. The reasons for these correlations are far from clear, especially in children and adolescents.

The main purpose of SLOPUS is to investigate the effects of reduced sleep on energy and substrate metabolism, and the relevant hormonal systems involved in the underlying mechanisms. Our hypothesis is that acute sleep deprivation in teenagers leads to increased hunger and desire to eat, increased spontaneous energy intake, decreased spontaneous physical activity, and increased fluctuation in the hormones that control energy metabolism.

The investigators aim to recruit twenty-four healthy, normal weight boys aged 15-19 years with normal sleep pat-terns. The study will be conducted as a randomized, crossover study with two conditions. Each participant will be subjected to short sleep (4 hours) and normal sleep (9 hours), in random order, for three consecutive nights in a respiration chamber. They will stay in the chamber for the 24 hours before the last night. In the respiration chamber energy turnover is measured - both how much energy and also the type of substrate combusted. The chamber is equipped with a bed, toilet, television, computer, and communication. Food and drink can be supplied via an airlock. Measurements in the chamber include volitional activities and sleep duration/quality.

Energy turnover will be measured using a ventilated hood system on the first and last day. Here the participants lie down on a bed with their heads under a transparent canopy for 25-minute intervals during the morning. Blood samples will also be taken during these periods. Meal tests will be served, where we measure the amount of food ingested, and subjects will be given questionnaires about hunger and satiety to fill out. Physical activity and heart rate will be measured throughout the trial.

Thus, the present study is likely to result in a number of new and important findings regarding the impact of impaired sleep on energy balance and it might improve the recommendations for optimal sleep in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* normal weight (5th percentile to less than the 85th percentile)

Exclusion Criteria:

* self-reported sleep problems (Pittsburgh Sleep Quality Index score >5);
* night work;
* variable sleep habits or habitual daytime naps;
* regular physical exercise (>3 hours/week);
* excessive intake of alcohol (>7 drinks/week);
* excessive intake of caffeine (>300 mg/day);
* smoking;
* substance abuse;
* use of prescription medications or over-the-counter drugs affecting sleep or metabolism;
* chronic diseases (e.g. cancer, asthma, back pain, thyroid disease, heart disease, diabetes, etc.)
* history of neurological, medical or sleep disorders;
* trans-meridian travelling the last month;
* eating disorder;
* irregular eating schedule (e.g. skipping breakfast);
* unable to comply with the protocol.

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | Over the course of 24 hours on day 3
  Energy expenditure and substrate oxidation rate will be assessed by 24-hour indirect whole-body calorimetry (respiration chamber) on the basis of measurements of oxygen consumption, carbon dioxide production, and nitrogen excretion in urine.

SECONDARY OUTCOMES:
Spontaneous energy intake | Measured after a maximum of 30 minutes meal time on day 1 and day 4
  In an attempt to measure spontaneous energy intake in an experimental context, the participant will be given an ad libitum lunch at noon. The ad libitum meal is a homogenous meal with a macronutrient composition of: 15 E%; fat: 30 E%; carbohydrate: 55 E%.The portion of pasta is larger than the expected participant's intake. The meal will be weighted before and after the lunch and ad libitum energy intake is assessed from the amount of the meal consumed by a food technician.
Spontaneous physical activity | 24 hours for 3 consecutive days
  Spontaneous physical activity is measured by a wrist worn actigrpahy device during the three days of intervention. Moreover, spontaneous activity in the respiration chamber will be assessed by in-biuld microwave radar detectors
Appetite regulating hormones and stress hormones | Measured every half hour over the course of 4 hours on day 1 and day 4
  Hormones are sampled from blood, saliva, and urine.
Hunger and desire to eat | Measured every hour or half hour over the course of 9 hours on day 1 and day 4
  Hunger and desire to eat is measured using visual analogue scales before and after a standardized breakfast meal challange and before and after an ad libitum meal.
Stress hormone (cortisol) | Measured at 7 am and 7.30 am on day 1 and day 4
  Hormones are sampled saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MD, PhD, Principal Investigator — Department of Human Nutrition, Faculty of LIFE Sciences, University of Copenhagen; Anders M Sjödin, MD, PhD, Principal Investigator — Department of Human Nutrition, Faculty of LIFE Sciences, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of LIFE Sciences, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Klingenberg L, Chaput JP, Holmback U, Jennum P, Astrup A, Sjodin A. Sleep restriction is not associated with a positive energy balance in adolescent boys. Am J Clin Nutr. 2012 Aug;96(2):240-8. doi: 10.3945/ajcn.112.038638. Epub 2012 Jul 3. PMID 22760574
- See also: Danish website — http://foodoflife.dk/slopus/